CLINICAL TRIAL: NCT05540379
Title: Role of Virtual Reality Simulators in Basic Hysteroscopy Training Competence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Hagar Elnashar
Record Dates: First submitted 2022-09-09; First posted 2022-09-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Hysteroscopy

STUDY DESIGN:
Intervention Model Description: the efficacy of VR simulator training in improving basic gynecological hysteroscopic skills
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Ob/Gyn physicians (Active Comparator): It is about 51 participants whom had performed less than 50 diagnostic hysteroscopies and hysteroscopic polypectomy.
  Interventions: Device: Virtual Reality Training
- Group B: Ob/Gyn physicians (Active Comparator): It is about 51 participants whom had performed at least 50 diagnostic hysteroscopies and hysteroscopic polypectomy.
  Interventions: Device: Virtual Reality Training

INTERVENTIONS:
Device: Virtual Reality Training — Training the obstetrics and Gynecologist Residents on Virtual endoscopic simulation and skills acquisition

SUMMARY:
Evaluation the efficacy of Virtual Reality simulator training in improving basic gynecological hysteroscopic skills and assess training levels in Ob/Gyn residents, as compared to others with previous hysteroscopic experience.

DETAILED DESCRIPTION:
Diagnostic or operative hysteroscopy is one of the most common surgical intervention in gynecological surgery. In recent years, it has acquired a central role in diagnosis and treatment of a variety of uterine pathologies like fibroids, polyps and uterine malformations It is also pivotal in the management of primary or secondary infertility. Biopsy specimens are also sampled with hysteroscopy in the diagnosis of endometrial cancer.

In recent years, the technological advancements such as the use of small diameter (3,5mm) rigid hysteroscopes combined with "no touch" techniques have made hysteroscopy a commonly accepted procedure .

As a minimally invasive procedure, hysteroscopy is associated with fewer complications than traditional open surgery However, it is challenging to gain manual dexterity in hysteroscopy because of the fulcrum effect and the orientation between the two-dimensional screen and the three-dimensional uterine cavity. Other difficulties are the diminished tactile feedback and limited degrees of freedom, . Lack of proficiency in hysteroscopy can compromise patient safety by causing uterine perforation and trauma to neighboring organs. Also, pulmonary air embolisms and pulmonary edema are potential life-threatening complications.

Today it is generally accepted that the traditional apprentice-tutor model is no longer valid for training all skills necessary in Gynecological surgery and more specifically endoscopic surgery This agreement is based on the recognition that, in contrast to open surgery, endoscopic surgery demands surgical skills and psychomotor skills that should not necessarily be trained simultaneously. Increasing evidence strongly suggests that psychomotor skills must be trained earlier and outside the operating room, and several models have been proposed for this aim

ELIGIBILITY:
Inclusion Criteria:

1. Residents, assistant lecturers, lecturers, associate professors and professors in Ob/Gyn department.
2. Group A: Ob/Gyn physicians who had performed less than 50 diagnostic hysteroscopies and hysteroscopic polypectomy.
3. Group B: Ob/Gyn physicians who had performed at least 50 diagnostic hysteroscopies and hysteroscopic polypectomy.

Exclusion Criteria:

1- Physicians who had previously attended VR simulator training course

Ages: 26 Years to 36 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Virtual Reality Training Score | from baseline to 6 months after the trainig
  • To compare the final score achieved by the physicians who had performed less than 50 diagnostic hysteroscopies and hysteroscopic polypectomy after 3 training sessions on VR hysteroscopy simulator with the score achieved by physicians who had performed at least 50 diagnostic hysteroscopies and hysteroscopic polypectomy to ensure the role of VR in training for hysteroscopic polypectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Fawzi El-Minawi, Professor, Study Chair — Department of obstetrics and gynecology, Faculty Of Medicine, Cairo University; Nadine A Sherif, Professor, Principal Investigator — Department of obstetrics and gynecology, Faculty Of Medicine, Cairo University
Locations (1):
- Faculty of Medicine - Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided